CLINICAL TRIAL: NCT02622048
Title: STAGE 1: Investigating Attributions and Expressed Emotion in Parents With and Without Psychosis STAGE 2: Investigating the Use of a Self-directed Parenting Programme With Parents Experiencing Psychosis
Brief Title: Understanding and Helping Families: Parents With Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lauren Stockton, PhD Clinical Psychology Student, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15209: 15/NW/0532
Record Dates: First submitted 2015-11-20; First posted 2015-12-04 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Parenting; Psychosis; Schizophrenia
Keywords: Mental Health; Psychosis; Parent
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stage 2 Parents experiencing psychosis (Experimental): Parents all receive the self-directed Triple P Positive Parenting Programme
  Interventions: Behavioral: Triple P Positive Parenting Programme

INTERVENTIONS:
Behavioral: Triple P Positive Parenting Programme — 10 week self-directed (guided) parenting intervention promoting self-belief, parenting confidence/self-efficacy and problem solving skills.

SUMMARY:
The purpose of this trial is to explore parent-child interactions in parents with and without psychosis, and ascertain whether a brief (10 week) supported self-help parenting program offered to parents in their own homes can help improve parents' self-efficacy and general well-being, as well as interpretations of their parent-child relationship and child behaviour in children who are 3-10 years old.

DETAILED DESCRIPTION:
The trial will be split into two stages.

Stage 1: Parents with no history of serious mental health problems and parents who have a history of psychosis or schizophrenia, who have children aged 3-10 years old, will take part in the Revised Five Minute Speech Sample (FMSS) and the Modified Camberwell Family Interview (CFI). They will also complete various measures looking at parental well-being, depression, anxiety and stress as well as parenting behaviours and interpretations of their child behaviour. In addition the PANSS interview will also be used. These interviews will be coded to investigate attributional patterns.

Stage 2: Parents who are experiencing psychosis, who took part in stage 1 will proceed to stage 2 if they want to. Parents will be seen weekly and take part in a guided self-help parenting intervention. This will require weekly visits over 10 weeks to the parents. During this time, symptoms, mood, general well-being and parenting behaviours will be monitored.

There will be no randomisation: all parents experiencing psychosis will receive the intervention.

Children do not attend the sessions, but it is hoped that parents practice the skills learned.

ELIGIBILITY:
Inclusion Criteria for parents with psychotic illnesses

1. Presence of ICD-10 schizophrenia-spectrum diagnosis (F20-29).
2. Primary parental caregiver for index child. This includes 10 hours of contact time with their child.
3. Over 18 years of age.
4. Have at least one child aged 3-10 years old.
5. Identify difficulties in parenting during assessment.
6. Proficient in written and spoken English.
7. Capacity to provide informed consent.

Exclusion Criteria for parents with psychotic illnesses

1. Parents with a schizophrenia-spectrum diagnosis who have recently been discharged from acute in-patient care, and have less than four weeks of stabilisation. This will enable the individual sufficient time to readjust to living in the community and ensure symptom stabilisation before taking part in a study.
2. Parents who have no regular contact with the index child or where there is known intention for their child to be removed.
3. Parents who present with child protection of safeguarding issues.
4. Parents seeking or receiving support from services regarding child management issues.
5. Parents actively involved in other structured programmes.

Inclusion Criteria matched comparison group of parents for stage 1

The comparison group of parents will be matched for age, education, socioeconomic status and family composition where possible

1. No previous history of psychotic illnesses.
2. Primary parental caregiver for index child. This includes 10 hours of contact time with their child.
3. Over 18 years of age.
4. Have at least one child aged 3-10 years old.
5. Identify difficulties in parenting during assessment.
6. Proficient in written and spoken English.
7. Capacity to provide informed consent.

Exclusion Criteria for comparison group

1. Parents with schizophrenia-spectrum symptoms, diagnosis or history.
2. Parents who have no regular contact with the index child or where there is known intention for their child to be removed.
3. Parents seeking support from services regarding child management issues.
4. Parents actively involved in other structured programmes.
5. Parents/caregivers who do not have good working knowledge of English. They should have enough practical experience to be able to adequately use the English language to understand and respond to questions and to read and complete questionnaires.
6. Insufficient language or cognitive ability to participant fully or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Initial Ax, Multiple Baseline Ax, Final Baseline Ax, 10 support sessions Ax, End Ax, Follow Up Ax. Ax from 0 - 16 weeks with 3 and 6 month follow up
  Assessment of parental symptoms, mood, behaviours, aswell as social performance and depression
Five Minute Speech Sample (FMSS) | Initial Ax, End Ax, Follow up Ax. Ax from 0 - 16 weeks with 3 and 6 month follow up
  Assessment of Expressed Emotion using a 5 minute uninterrupted interview
Modified Camberwell Family Interview (CFI) | Initial Ax only
  In depth assessment of Expressed Emotion using a modified version of the CFI. This version is for parents of well children.

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21) | Initial Ax, Multiple Baseline Ax, Final Baseline Ax, 10 support sessions Ax, End Ax, Follow Up Ax. Ax from 0 - 16 weeks with 3 and 6 month follow up
  Self-reported depression, anxiety and stress using a short form scale
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Initial Ax, Final Baseline Ax, End Ax, Follow Up Ax. Ax from 0 - 16 weeks with 3 and 6 month follow up
  Self-reported general well-being
Eyberg Child Behaviour Inventory (ECBI) | Initial Ax, Final Baseline Ax, 10 support sessions Ax, End Ax, Follow Up Ax. Ax from 0 - 16 weeks with 3 and 6 month follow up
  Parents self-reported child problem behaviour
Strengths and Difficulties Questionnaire (SDQ) | Initial Ax, Final Baseline Ax, End Ax, Follow Up Ax. Ax from 0 - 16 weeks with 3 and 6 month follow up
  Parents self-reported child behaviour assessing different aspects of behaviour, e.g.,: emotional symptoms, conduct problems, hyperactivity/inattention.
Parenting and Family Adjustment Scale (PAFAS) | Baseline, 1, 5, 10, follow up
  An assessment of parenting skills and family relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Stockton, Principal Investigator — The University of Manchester
Locations (1):
- The University of Manchester, Manchester, Lancashire, United Kingdom